

# APL-B-022-15 (NCT03117361)

A Phase II Trial of Plitidepsin (Aplidin®) in Combination with Bortezomib and Dexamethasone in Multiple Myeloma Patients Double Refractory to Bortezomib and Lenalidomide

STATISTICAL ANALYSIS PLAN

Version: 1.0

Date: 13-December-2016

### TABLE OF CONTENTS

| 1 | ST | UDY RATIONALE | 6 |
|---|---|---|---|
| 2 | ST | UDY DESIGN | 6 |
| 3 | OB | BJECTIVES AND ENDPOINTS | 7 |
| | 3.1 | Primary Objective | 7 |
| | 3.2 | Secondary Objectives | 7 |
| | | Endpoints | 7 |
| 4 | PA | TIENTS EVALUABILITY CRITERIA | 8 |
| | 4.1 | Definition of Patient Sets for Analysis | 8 |
| 5 | SA | MPLE CONSIDERATIONS | 8 |
| 6 | ST | ATISTICAL METHODOLOGY FOR EFFICACY | 9 |
| | 6.1 | Planned Analyses and Definitions | 9 |
| | 6.1 | .1 Primary Endpoint | 9 |
| | 6.1 | .2 Secondary Endpoints | 9 |
| | | .3 Other Definitions | 9 |
| | 6.2 | Efficacy Analysis Methods | 10 |
| | | .1 Primary Analysis | 10 |
| | | .2 Secondary Analyses | 10 |
| | 6.2 | .3 Other Exploratory Analyses | 10 |
| 7 | ST | ATISTICAL METHODOLOGY FOR SAFETY | 10 |
| | 7.1 | Adverse Events | 10 |
| | 7.2 | Clinical Laboratory Evaluation | 11 |
| | 7.3 | Vital Signs, Physical Examination, Left Ventricular Ejection Fraction (LV | /EF) and |
| | | rocardiogram Findings | 12 |
| | 7.4 | Deaths and Other Serious Adverse Events | 12 |
| 8 | OT | HER ANALYSES | 12 |
| | 8.1 | Baseline and Demographic Data | 12 |
| | 8.2 | Treatment Administration | 12 |
| | 8.3 | Subsequent Therapy | 13 |
| | 8.4 | Protocol Deviations | 13 |
| | 8.5 | Pharmacokinetic and Pharmacodynamic Analyses | 13 |
| | 8.6 | Pharmacogenomic Analyses | 13 |
| | 8.7 | Decimal Places | 13 |
| | 8.8 | Imputation of Incomplete Dates | 13 |
| | 8.9 | Subgroup Analyses | 14 |
| | 8.10 | Methods for Handling Missing Data | 14 |
| | 8.11 | Interim and Group Sequential Analyses | 14 |
| | 8.12 | Data Analysis Conventions | 14 |
| 9 | ST | ATISTICAL SOFTWARE | 14 |
| | <u>APPE</u> | ENDIX I | 15 |
| 1( | ) Stu | ndy Patients | 15 |
| | 10.1 | Patient Disposition | 15 |
| | 10.2 | Reasons for Treatment and Study Discontinuation | 16 |
| | 10.3 | Protocol Deviations | 17 |

| 11 | Efficacy | / Evaluation | 17 |
|---|---|---|---|
| 1 | 1.1 | Demographic and Other Baseline Characteristics | 17 |
| | 11.1.1 | Patient Characteristics at Baseline | 17 |
| | 11.1.2 | Disease at Diagnosis, Time from Diagnosis and Current Disease | 18 |
| | 11.1.3 | Cytogenetics | 19 |
| | 11.1.4 | Prior Anticancer Therapy | 19 |
| | 11.1.5 | Physical Examination, Vital Signs, Electrocardiogram and Other Tests | 20 |
| | | Viral Serology | 22 |
| | 11.1.7 | Hematological Values at Baseline | 23 |
| | 11.1.8 | Biochemical Values at Baseline | 23 |
| | 11.1.9 | Other Metabolic Values at Baseline | 24 |
| | 11.1.10 | Signs and Symptoms at Baseline | 24 |
| | <u>11.1.11</u> | Concomitant Medication/Procedures at Baseline | 24 |
| 1 | 1.2 | Efficacy Analysis | 25 |
| | 11.2.1 | Primary Analysis | 25 |
| | 11.2.2 | Secondary Analyses | 25 |
| | 11.2.3 | Other Exploratory Analyses | 26 |
| | 11.2.4 | Characteristics of Responders | 27 |
| | 11.2.5 | Multivariate analyses | 27 |
| <u>12</u> | Safety A | Analysis | 29 |
| <u>12</u> | 2.1 | Extent of Exposure | 29 |
| | 12.1.1 | Treatment Administration | 29 |
| | 12.1.2 | Cycle Delays | 29 |
| | 12.1.3 | Dose Omissions | 31 |
| | 12.1.4 | Dose Reductions | 31 |
| <u>12</u> | 2.2 | Adverse Events (AEs) | 32 |
| | 12.2.1 | Display of Adverse Events | 32 |
| <u>12</u> | 2.3 | Serious Adverse Events and deaths. | 35 |
| | 12.3.1 | Serious Adverse Events | 35 |
| | 12.3.2 | <u>Deaths</u> | 36 |
| <u>12</u> | 2.4 | Clinical laboratory evaluation | 37 |
| | 12.4.1 | Hematological Abnormalities | 37 |
| | 12.4.2 | Biochemical Abnormalities | 38 |
| | 12.4.3 | Other metabolic parameters | 39 |
| | 12.4.4 | Laboratory values over time | 39 |
| <u>12</u> | 2.5 | Vital Signs, Physical Findings, LVEF, ECG and Other Tests Related to S | afety |
| | | 41 | |
| | 12.5.1 | Vital Signs and Physical Findings | 41 |
| | 12.5.2 | LVEF and ECG | 42 |
| 12 | 2.6 | Concomitant Medication / Procedures according to the ATC Classification | <u>n. 42</u> |
| _ | 2.7 | Safety Analysis in Special Subgroups. | 43 |
| _ | 2.8 | MM Serum/Urine Protein Measurements | 44 |
| 13 | DB List | ings | 45 |
| 14 | ICH Lis | tings | 46 |

### LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

**AE(s)** Adverse Event(s)

ALT Alanine Aminotransferase AP Alkaline Phosphatase

**ASCT** Autologous Stem Cell Transplantation

**AST** Aspartate Aminotransferase

ATC Anatomical Therapeutic Chemical

**ATC-WHO** Anatomical Therapeutic Chemical Drug Classification by the

World Health Organization

BM Bone Marrow
BSA Body Surface Area
CBR Clinical Benefit Rate
CI Confidence Interval
CMV Cytomegalovirus

**CPK** Creatine Phosphokinase

**CPK-MB** Serum CPK Isoenzymes (Found In Cardiac Muscle)

CR Complete Response
CrCl Creatinine Clearance
CRF Case Report Form

CTCAE Common Terminology Criteria for Adverse Events

**D** Day

**DB** Data Base

DLT Dose Limiting Toxicity
 DOR Duration of Response
 ECG Electrocardiogram
 ECHO Echocardiogram

**ECOG PS** Eastern Cooperative Oncology Group Performance Status

**e-CRF** Electronic Case Report Form

**EFS** Event-free Survival **EOT** End-of-treatment

**G-CSF** Granulocyte Colony Stimulating Factor

**GGT** y-glutamyl Transpeptidase

H Hour

**HBV** Hepatitis B virus

**HCG** Human Chorionic Gonadotropin

**HCV** Hepatitis C virus

**HDT** High Dose Chemotherapy

HIV Human Immunodeficiency Virus

HLA Human Leukocyte Antigen
Hematonoietia Stem Cell Tr

HSCT Hematopoietic Stem Cell Transplantation
ICH International Conference on Harmonization
IMWG International Myeloma Working Group

Ig Immunoglobulin


**IMIDs** Immunomodulatory Drugs

IMP Investigational Medicinal Product ISS International Staging System

i.v Intravenous

**LDH** Lactate Dehydrogenase

**LVEF** Left Ventricular Ejection Fraction

**MedDRA AE** Medical Dictionary for Regulatory Activities for Adverse Events

MM Multiple Myeloma
MOA Mechanism of action
MR Minimal Response

MUGA scan Multiple Uptake Gated Acquisition Scan

NA Not Applicable

NCI-CTCAE National Cancer Institute Common Toxicity Criteria

NOS Not Otherwise Specified ORR Objective Response Rate

OS Overall Survival

OS6 Overall Survival Rate at 6 Months
OS12 Overall Survival Rate at 12 Months

**PCR** Polymerase Chain Reaction

PD Progressive Disease
PDy Pharmacodynamics
PFS Progression-free Survival
PGx Pharmacogenomics
PI Proteasome Inhibitor
PK Pharmacokinetics
PN Peripheral Neuropathy
PD Progressive Disease
Pharmacodynamics
Progressive Disease
Progression-free Survival
Progre

PR Partial Response
PS Performance Status

**R-ISS** Revised International Staging System

**RR** Response Rate

SAE(s) Serious Adverse Event(s)

s.c. Subcutaneous

**sCR** Stringent Complete Response

**SD** Stable Disease

SFLC Serum Free Light Chains
SOC System Organ Class
StD Standard Deviation
TTP Time To Progression

VGPR Very Good Partial Response

**WBC** White Blood Cells

wk Week(s)

**WOCBP** Woman/Women of Childbearing Potential

### 1 STUDY RATIONALE

- Multiple myeloma (MM) is a malignant plasma-cell disorder characterized by the production of a monoclonal protein from plasma cells in the bone marrow (BM).
- In the Western hemisphere, about 1% of cancer-related deaths are due to myeloma.
- MM is still an incurable disease. As front-line treatment to reduce tumor burden, hematopoietic stem cell transplantation (HSCT) as well as emergent drugs used in newly diagnosed patients offer the best chance for long-term survival. However, while many studies have shown the benefits of this approach, most patients will relapse. Thus, additional therapeutic options are needed for these patients.

A full rationale for the study design including the choice of the double refractory patient population and the use of the combination of plitidepsin with bortezomib and dexamethasone may be found in the appropriate sections of the study clinical protocol (section 1.5).

### 2 STUDY DESIGN

This is a multi-center, open-label, single arm, non-comparative phase II trial, designed to evaluate the efficacy of plitidepsin in combination with bortezomib and dexamethasone in patients with MM double refractory to bortezomib and lenalidomide. Plitidepsin will be administered as a 3-hour (h) i.v. infusion at a dose of 5 mg/m², on Day (D) 1 and 15, q4wk, bortezomib will be administered as a s.c. injection at a dose of 1.3 mg/m² on D1, 4, 8 and 11, q4wk and dexamethasone will be taken orally at a dose of 40 mg/day on D1, 8, 15 and 22, q4wk.

Patients will be evaluated at scheduled visits in three trial periods: pre-treatment, treatment and follow-up.

The **pre-treatment period** includes screening and baseline visits. Baseline assessment consists of a detailed history of pre-existing diseases, physical examination and clinical neurological assessment, ECOG PS, ECG, LVEF and laboratory tests, urinalysis, hepatitis B and C virus screening and serum pregnancy tests for WOCBP.

During the **treatment period**, all patients are to attend trial center visits on Day 1, 4, 8, 11 and 15 on an every four-week basis to assess safety and toxicity. All patients are to attend an end-of-treatment (EOT) visit 30 ( $\pm$ 5) days after the last dose of trial therapy.

A cycle is defined as 28 days, plus any additional days required for dosing delays due to any reason.

After completion of the treatment period or in case of discontinuation, patients are to attend **follow-up visits**. Patients will be followed for AEs during 30 days after the last administration of trial drug and until their resolution. In addition, patients will be followed every three months to assess disease status.

A full description for the study may be found in the appropriate sections of the study clinical protocol.

### 3 OBJECTIVES AND ENDPOINTS

### 3.1 Primary Objective

• To evaluate the efficacy of plitidepsin in combination with bortezomib and dexamethasone in patients with MM double refractory to bortezomib and lenalidomide in terms of overall response rate (ORR), including stringent complete response (sCR), complete response (CR), very good partial response (VGPR) and partial response (PR).

### 3.2 Secondary Objectives

- To evaluate time-to-event efficacy endpoints of plitidepsin in combination with bortezomib and dexamethasone, i.e., duration of response (DOR), time to progression (TTP), progression-free survival (PFS) and event-free survival (EFS).
- To evaluate overall survival (OS) and OS rate at 6 and 12 months (OS6 and OS12, respectively).
- To evaluate the safety and tolerability of plitidepsin in combination with bortezomib and dexamethasone.
- To study the pharmacokinetics (PK) and pharmacodynamics (PDy) of plitidepsin in combination with bortezomib and dexamethasone.
- To obtain pharmacogenomic information (Pharmacogenomics [PGx]) on markers of response to plitidepsin and bortezomib treatment.

### 3.3 Endpoints

### **Primary endpoint:**

 ORR, defined as the percentage of patients with sCR, CR, VGPR or PR according to IMWG response criteria.

### Secondary endpoints:

- DOR, defined as the time from the first observation of response to the time of PD, with censoring of deaths due to causes other than PD
- TTP, defined as the time from the date of first drug administration to the date of PD.
- PFS, defined as the time from the date of first drug administration to the date of PD or death (of any cause).
- EFS, defined as the time from the date of first drug administration to the date of drugrelated events leading to treatment discontinuation, PD or death (of any cause), whichever comes first.
- OS, defined as the time from the date of the first dose to the date of death or last patient contact.
- OS6 / OS12, defined as the Kaplan-Meier estimate of the percentage of patients who are alive at six/twelve months after first drug administration.

Treatment safety [AEs, SAEs and laboratory abnormalities] graded according to the NCI-CTCAE, v. 4. Dose reductions, skipped doses or dose delays required due to treatment-related AEs, and reasons for treatment discontinuations will be analyzed. Other supportive exploratory endpoints are defined in section 6.1.3.

### 4 PATIENTS EVALUABILITY CRITERIA

The study population will include patients with MM double refractory to bortezomib and lenalidomide. To be enrolled in this study, the patients must meet all inclusion criteria and no exclusion criteria.

### 4.1 Definition of Patient Sets for Analysis

"All Included Patients" analysis set is defined as all patients who are included in the study (excluding screening failures), independent of whether they received the study drug.

"All Evaluable for Safety Patients" analysis set is defined as all included patients who receive at least part of one dose or infusion of plitidepsin.

"All Evaluable for Efficacy Patients" analysis set is defined as all included patients who receive at least one complete treatment cycle (two plitidepsin infusions, four bortezomib injections, four doses of dexamethasone), or the equivalent doses over two cycles and must have had at least one disease assessment.

"All Responder Patients" analysis set is defined as all evaluable patients for efficacy who have partial response or better as overall best response.

#### 5 SAMPLE CONSIDERATIONS

Patients will be treated to test the null hypothesis  $(H_0)$  that 20% or fewer patients achieve a response according to IMWG criteria  $(p \le 0.20)$  versus the alternative hypothesis  $(H_1)$  that 40% or more patients achieve a response according to IMWG criteria  $(p \ge 0.40)$ . The variance of the standardized test will be based on the empirical estimate. The type I error rate (alpha) associated with this one-sided test is 0.025 and the type II error rate (beta) is 0.1; hence, statistical power is 90%. In order to test these hypotheses, it is necessary to recruit 64 evaluable patients.

A futility analysis based on the primary endpoint (ORR) is planned for the time when the first 20 evaluable patients have been recruited. The futility analysis will commence once patient number 20 has completed two full treatment cycles. Patient recruitment will not be halted during the conduct of this futility analysis. A spending function defined by the Gamma family with parameter (-2) has been selected. If there are two or fewer responders according to boundaries and sample size assumptions, then the alternative hypothesis could be rejected and recruitment might be stopped at that time. Otherwise, patient accrual will continue to a total of 64 patients.

Overall, if  $\geq$  21 (i.e., 33%) patients achieve a response, then the null hypothesis can be rejected.

### 6 STATISTICAL METHODOLOGY FOR EFFICACY

### 6.1 Planned Analyses and Definitions

Frequency tables will be performed for categorical variables, whereas continuous variables will be described by means of summary tables that will include the mean, standard deviation (StD), median, minimum, and maximum of each variable.

The "All Evaluable for Efficacy Patients" analysis set will be used for the analyses of ORR, TTP, PFS, EFS, OS, clinical benefit rate (CBR) and disease control rate (DCR).

The "All Responder Patients" analysis set will be used for the analyses of the DOR and time to response.

### 6.1.1 Primary Endpoint

The *ORR* is calculated as the percentage of the number of responders, based on the IMWG response criteria, divided by the total number of patients.

### 6.1.2 Secondary Endpoints

The **DOR** will be analyzed for all patients in whom a response has been observed and is defined as the time, in months, from the date of first documentation of response to the date of disease progression. Response will be assessed according to the IMWG classification response criteria. Deaths due to causes other than PD will be censored.

**TTP** is defined as the time, in months, from the date of the first infusion to the date of documented PD or death due to PD. TTP will be censored on the date of the last tumor assessment or on the date of the first drug administration if there are no tumor assessments.

**PFS** is defined as the time, in months, from the date of first drug administration to the date of documented PD, or death (of any cause). If any patient is lost to follow-up before PD or receives another antitumor therapy, PFS will be censored on the date of the last tumor assessment. If there are no tumor assessments, these parameters will be censored on the date of the first drug administration.

**EFS** is defined as the time, in months, from the date of first drug administration to the date of onset of the first drug-related event leading to treatment discontinuation, documented PD or death. The censoring rules defined above for PFS will be used for EFS.

**OS**, defined as the time, in months, from the date of first drug administration to the date of death (of any cause) or last patient contact (in this case, survival will be censored on that date).

*OS6/OS12*, defined as the Kaplan-Meier estimate of the percentage of patients who are alive at six/twelve months after first drug administration.

### 6.1.3 Other Definitions

**CBR** was defined in the protocol as SD or better but to homogenize with nowadays standard practice it has been considered to report it as MR or better. Nevertheless, to maintain the definition in the protocol, it will be called **DCR** for the analyses and it is defined as SD or better.

**Duration of Minor Response,** defined as the time, in months, from the first observation of MR to the time of PD, with censoring of deaths due to causes other than PD.

*Time to response,* defined as the time, in months, from the first drug administration to the first documentation of response.

### 6.2 Efficacy Analysis Methods

### 6.2.1 Primary Analysis

For the evaluation of the primary endpoint, *ORR*, the exact binomial estimator (count and percentage) including its 95% confidence interval will be used.

### 6.2.2 Secondary Analyses

Time-to-event variables (DOR, TTP, PFS, EFS and OS) and their fixed time estimates (i.e. OS6 and OS12) will be analyzed according to the Kaplan-Meier method.

Multivariate analyses by logistic regression could be carried out for ORR, and Cox regression for time-to-event endpoints, as supportive analysis.

If appropriate, exploratory multivariate models (e.g. Logistic/Cox regression) will include prognostic factors/covariates widely reported and recognized by hematologist such as: sex, age at diagnosis, baseline ECOG, Body Surface Area, MM type, number of prior lines of anti-myeloma treatment, previous SCT, cytogenetics and/or other covariates according to the hematologist's criteria.

### 6.2.3 Other Exploratory Analyses

The CBR is calculated as patients with sCR, CR, VGPR, PR, MR divided by the number of patients. The DCR is calculated as patients with sCR, CR, VGPR, PR, MR or SD divided by the number of patients.

Duration of minor response and time to response will be analyzed according to the Kaplan-Meier method.

Waterfall plot will be used to describe the maximum reduction of M-protein in serum and urine.

#### 7 STATISTICAL METHODOLOGY FOR SAFETY

The analysis of the secondary endpoint treatment safety will be based on the "All Evaluable for Safety Patients" analysis set.

### 7.1 Adverse Events

All the adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

The adverse event evaluation will be coded with the National Cancer Institute-Common Toxicity Criteria (NCI-CTC), version 4.

As far as all the adverse events are concerned, the NCI-CTC grade will be used wherever an NCI-CTC grading exists. Otherwise, the severity will be noted. As a convention, the term «Grade» will always be used. Adverse events will be described according to the worst NCI-CTC grade or, for events which do not form the subject of NCI-CTC classification, according to the worst severity.

AEs reported in EOT visit will be imputed to last cycle.

An overall summary of adverse events will be done by body system and preferred term, by severity (worst toxicity grade), by relationship to the study drug/s (drug related or relationship unknown / all adverse events regardless of relationship), and by AE outcome. Only events reported by the Investigator as 'not related to plitidepsin +/- bortezomib +/- dexamethasone' will be excluded from the trial analysis of drug-related events. A second set of tables including all events will also be presented, and a third set of tables including treatment emergent events will also be presented.

A frequency table will be made for the AEs leading to cycle delay, dose reduction, dose omission, or withdrawal of study medication. Adverse events with outcome of death will also be presented by relationship to the study drugs.

All events entered in Adverse Event form with the onset date before the first drug administration, will be reported as Signs and symptoms. Only those events with start date after or on the date of first infusion will be included in AE tables in Safety section (except those already present at baseline).

### 7.2 Clinical Laboratory Evaluation

Laboratory results will be classified according to the NCI-CTC version 4.

For hematology values: absolute neutrophil count, lymphocyte count, WBC count, platelet count and hemoglobin worst grade per patient and per cycle will be displayed.

Laboratory results reported during the EOT visit will be imputed to last cycle.

Overall cross tabulation will be used to present the worst grade during treatment versus the baseline toxicity grade for anemia, lymphopenia, leukopenia, neutropenia and thrombocytopenia, and also versus treatment-emergent events (i.e., those that worsened or appeared for the first time during treatment).

The worst grade per patient during treatment and per cycle will also be calculated for biochemical tests: ALT, AST, total bilirubin, AP, CPK, GGT, creatinine, calcium (corrected by albumin levels), potassium, sodium, magnesium, glucose and albumin.

Time and duration of AST, ALT and CPK increases, platelet count and neutrophil count in cycles with grade 3-4 abnormality will be tabulated.

Overall cross tabulation will be presented for the worst grade during treatment versus the baseline toxicity grade of AST, ALT, bilirubin, creatinine, AP, CPK and electrolytes; and also versus treatment-emergent events.

## 7.3 Vital Signs, Physical Examination, Left Ventricular Ejection Fraction (LVEF) and Electrocardiogram Findings

Tabulation will be used to summarize the performance status, body weight, and LVEF and electrocardiogram abnormalities at baseline and during the treatment, if appropriate, for each patient.

#### 7.4 Deaths and Other Serious Adverse Events

Deaths and Serious Adverse Events will be tabulated according to their relationship with the study treatment and time from last dose ( $\leq 30d / > 30d$ ).

#### 8 OTHER ANALYSES

Categorical variables will be described in frequency tables using counts and percentages. Continuous variables will be described by median, mean, standard deviation, minimum and maximum

### 8.1 Baseline and Demographic Data

Baseline data such as demographics, multiple myeloma history, prior therapy, prior relevant history, signs and symptoms, electrocardiogram, LVEF, laboratory values and concomitant medication (ATC-WHO coded) will be described following standard tables detailed in Appendix I. When two or more assessments have been done for the same parameter/test, the last assessment before or on the first drug administration will be taken into account for the analysis.

#### 8.2 Treatment Administration

Total cumulative dose, time on treatment, dose intensity and relative dose intensity, cycle delays, dose omissions and dose reductions will be described following standard tables detailed in Appendix I.

Total cumulative dose, is the sum of all the study drug doses from the first cycle until last cycle, including the dose received in the last cycle.

Patients will be considered to be on-treatment for the duration of their treatment and 30 days following the last treatment dose. If the patient starts any new antitumor therapy outside this clinical trial or dies within 30 days of last treatment dose, the date of administration of this new therapy or the date of death will be considered the date of treatment discontinuation.

However, as a convention, for dose intensity calculation purposes, the duration of the last cycle is considered to be 28 days.

Intended dose intensity is the planned dose per cycle divided by the planned number of weeks by cycle.

Absolute dose intensity is the actual cumulative dose divided by the number of weeks of treatment. Relative dose intensity (%) is the ratio of absolute dose intensity divided by the intended dose intensity.

The item «Infusion delayed/omitted: yes/no» in the case report form (CRF) will be used to calculate the delayed infusions. For cycles considered as delayed by the investigator, the delay will be calculated as:

Delay: Date of current drug administration – Date of previous drug administration – 28.

The first infusion of the first cycle will be excluded from all cycle delays and cycle modification calculations.

### 8.3 Subsequent Therapy

A table summarizing all subsequent therapies received after treatment discontinuation will be shown.

Time to first subsequent therapy or death will be analyzed as a measure of the time from first drug administration to treatment failure that leads to the need of a further treatment regimen.

#### 8.4 Protocol Deviations

Analysis of inclusion/exclusion criteria deviations, retreatment restrictions, used concomitant medication and clinically relevant discontinuations will be done as described in Appendix I.

### 8.5 Pharmacokinetic and Pharmacodynamic Analyses

These analyses will be detailed in separate documents.

### 8.6 Pharmacogenomic Analyses

This analysis will be detailed in a separate document.

#### 8.7 Decimal Places

By default, all results will be rounded to one decimal, except in the case where variables are integer; in that case, they will be reported without decimals, for example, age in years, number of sites. For representing p-values four decimals will be selected as default but they could be rounded to fewer decimals if necessary.

### 8.8 Imputation of Incomplete Dates

The dates of certain historical or current clinical activities are a key component of statistical analysis. Incomplete date appears when day, month or year is/are missing, and it can be imputed so that variables like time to and duration of a certain event can be calculated. When none day, month or year are available, then the date is missing, no imputation can be applied.

#### Before registration

If day of a date is unknown then the imputed day will be the 15<sup>th</sup> of the month, if the month is also unknown then the imputed date will be July 1st. This assumption will be valid if the imputed date is earlier than the registration date; otherwise the imputed date will be the first day of the registration month (i.e. 1/Month of registration date/Year).

#### Between treatment start and end of treatment

All date variables during treatment where information is needed and is not fully available, for example adverse events or concomitant medications, will be subject of imputation by means of SAS programming. If the day of a date is unknown then the imputed day will be 1, if the month is also unknown then the imputed date will 1/January. This assumption will be valid if the imputed date is earlier than the treatment start date; otherwise, the imputed date will be the treatment start date.

### After end of treatment

To ensure the most conservative approach for time-to-event variables (i.e. DOR, TTP, PFS, EFS and OS) that can be affected by missing values, the following rules will be implemented: if the day of a date is unknown then the imputed day will be the first of the month. This assumption will be valid if the imputed date occurs later than the last drug administration date; otherwise the imputed date will be the last drug administration date plus 1 day.

### 8.9 Subgroup Analyses

Specific subgroup analysis will be developed according to those variables considered clinically relevant.

The influence of prognostic factors on the efficacy endpoints will be studied in the multivariate analysis. These prognostic factors to be considered are; multiple myeloma status (relapse, refractory or relapse and refractory), cytogenetic risk (high risk vs standard risk), number of prior lines, etc.

Analysis of safety profile based on age, race, body mass index (BMI) or other clinically relevant variables will be performed.

### 8.10 Methods for Handling Missing Data

Missing values will not be included in the calculation of outputs.

### 8.11 Interim and Group Sequential Analyses

A futility analysis based on the primary endpoint (ORR) is planned for the time when the first 20 evaluable patients have been recruited. The analysis will commence once the last of the 20 patients has completed two full treatment cycles.

### 8.12 Data Analysis Conventions

All data analysis conventions, data calculations and grouping needed to perform the Clinical Study Report outside of this statistical analysis plan will be described in a separate document

### 9 STATISTICAL SOFTWARE

Medidata Rave® EDC will be used for data entry and clinical data management.

EAST v.6.3.1 has been used to calculate sample size.

SAS v.9.4 or superior will be used for all statistical analysis outputs.

#### APPENDIX I

All tables will be created at the time of each analysis planned in the protocol if applicable, and at study end.

Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate group size as appropriate.

If the number of categories or items does not yield appropriate tabular or graphic representations, detailed listings will be shown instead.

### 10 Study Patients

These analyses will be performed in "All Included patients" analysis set.

### 10.1 Patient Disposition

Main characteristics concerning inclusion in the study, withdrawal from the study and protocol deviations will be displayed in this section.

Table 10.1.1 Number of Patients Included, Evaluable for Safety, and Evaluable for the Main Endpoint.

| | N | % |
|-------------------------------------|---|---|
| All Included patients | | |
| All evaluable patients for safety | | |
| All evaluable patients for efficacy | | |

Listing 10.1.2 Patients who do not meet All Inclusion Criteria.

| Patient id. | Criterion number(s) and description |
|-------------|-------------------------------------|

Listing 10.1.3 Patients who meet Any Exclusion Criteria.

| Patient id. | Criterion number(s) and description |
|-------------|-------------------------------------|

Listing 10.1.4 Patients not Evaluable for Efficacy

| <u> </u> | J |
|-------------|--------|
| Patient id. | Reason |

Listing 10.1.5 Patient not Evaluable for Safety.

| Eleting 10:1.5 1 attent not Evaluate for Surety. | |
|--------------------------------------------------|--------|
| Patient id. | Reason |

Table 10.1.6 Patients Accrual by Institution

| | Country | Institution | N | % |
|--------------|-----------|---------------|---|---|
| | | Institution 1 | | |
| | Country 1 | | | |
| | | Total | | |
| | | Institution 1 | | |
| No. included | | | | |
| | | Total | | |
| | | Institution 1 | | |
| | Total | | | |
| | | Total | | |
| | | Institution 1 | | |
| | Country 1 | | | |
| | | Total | | |
| | | Institution 1 | | |
| No. treated | | | | |
| | | Total | | |
| | | Institution 1 | | |
| | Total | | | |
| | | Total | | |

### Table 10.1.7 Study Dates

| Date of first registration |
|-----------------------------------------|
| Date of first dose of the first patient |
| Date of last registration |
| Date of first dose of the last patient |
| Date of last dose |
| Date of last follow-up* |

<sup>(\*)</sup> Last follow-up or exam or procedure before clinical cut-off or study closure

### 10.2 Reasons for Treatment and Study Discontinuation

Table 10.2.1 Treatment Discontinuation

| | N | % |
|-------------------------------------------|---|---|
| Progressive disease | | |
| Treatment related adverse event | | |
| Non treatment related adverse event | | |
| Patient refusal to treatment | | |
| Investigator decision | | |
| Death | | |
| Other * | | |
| Total | | |
| N. ( 11 11 11 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | |

Note: This table will be based on treated patients .Other (\*) Specify (see listing 10.2.2)

### Listing 10.2.2 Reasons for Treatment Discontinuation Other than Progressive Disease.

| Patient id. | Reason | Last cycle | Comments |
|-------------|--------|------------|----------|

Note: This table will be based on treated patients

### Listing 10.2.3 Treatment Discontinuation due to AEs

| Patient id. | Cycle | Preferred<br>term code | Adverse event reported (verbatim) | Grade | Relationship | Onset date | Resolved<br>date | Seriousness<br>criteria | Outcome |
|---|---|---|---|---|---|---|---|---|---|

Note: This table will be based on treated patients

### Table 10.2.4 Study Discontinuation

| • | N | 0/0 |
|--------------------------------------|---|-----|
| Study termination (clinical cut-off) | | |
| Patient's refusal | | |
| Never treated | | |
| Death | | |
| Patient's follow-up completed | | |
| Lost to follow-up | | |
| Other * | | |
| Total | | |

Other (\*) See Listing 10.2.5

Listing 10.2.5 Study Discontinuation due to Other Reason

| Patient id. | Reason | Specify |
|-------------|--------|---------|

#### 10.3 Protocol Deviations

Listing 10.3.1 Protocol Deviations

| Patient id. | Deviation type | Description |
|-------------|----------------|-------------|

### 11 Efficacy Evaluation

### 11.1 Demographic and Other Baseline Characteristics

These analyses will be performed in "All Included patients" analysis set.

### 11.1.1 Patient Characteristics at Baseline

### Table 11.1.1.1 Baseline characteristics: Sex

| | N | % |
|--------|---|------|
| Male | X | XX.X |
| Female | | |
| Total | | |

Table 11.1.1.2 Baseline characteristics: Age at treatment registration

| N | Median | Mean | StD | Min | Max |
|---|--------|------|-----|-----|-----|

Table 11.1.1.3 Baseline characteristics: Age grouped

| | N | % |
|------------|---|------|
| <65 years | X | XX.X |
| 65-75 yeas | | |
| ≥75 | | |
| Total | | |

### Table 11.1.1.4 Baseline characteristics: Race

| | N | % |
|-------|---|------|
| White | X | XX.X |

| Total | | | | | | | |
|---|---|---|---|---|---|---|---|
| 11.1.2 Disea | ise at Diagno | sis, Time fro | m Diagnosis | s and C | urrent Di | isease | |
| Table 11.1.2.1 | Time from d | iagnosis to fi | rst infusion ( | months | ) | | |
| N | Median | Mean | StD | | Min | | Max |
| Table 11.1.2.2 | Time from la | ast PD to first | infusion (w | eeks) | | | |
| N | Median | Mean | StD | | Min | | Max |
| Table 11.1.2.3 | Multiple My | eloma Type. | | - IN | | % | |
| Secretory | | | | N<br>X | | XX.X | 7 |
| Oligosecretory | | | | 71 | | 7121,2 | <u> </u> |
| Non-Secretory | | | | | | | |
| Total | | | | | | | |
| Table 11.1.2.4 | Ig abnormal | ity at diagnos | is (for secret | ory and | oligosec | | IM). |
| | | | | N | | % | |
| IgG | | | | X | | XX.X | |
| IgA | | | | | | | |
| IgD | | | | | | | |
| IgE | | | | | | | |
| IgM | | | | | | | |
| Kappa light-chain D | | | | | | | |
| Lambda light-chain | Disease | | | | | | |
| Total | | | | | | | |
| Table 11.1.2.5 | Durie-Salmo | on Stage at Fi | rst Diagnosi | | | | |
| TA | | | | N | | %<br>XXX | , |
| IA | | | | X | | XX.X | |
| IB | | | | | | | |
| IIA | | | | | | | |
| IIB | | | | | | | |
| IIIA | | | | | | | |
| IIIB | | | | | | | |
| Total | | | | | | | |
| Table 11.1.2.6 | ISS Stage at | First Diagnos | sis. | | | | |
| T | | | | N | | %<br>XX X | , |
| I | | | | X | | XX.X | <u> </u> |
| II | | | | 1 | | | |
| Ш | | | | | | | |
| Not Done | | | | 1 | | | |
| Total | | | | | | | |
| Table 11.1.2.7 | Karyotype a | nd FISH at Fi | rst Diagnosi | S. | | | |
| | | | | N | | % | |
| Done | | | | X | | XX.X | <u> </u> |
| Not Done | | | | | | | |


| Total |
|-------|

Table 11.1.2.8 R-ISS Stage at Study Entry

| | N | % |
|------------------------------------------------------------------|---|------|
| I (ISS stage I and standard-risk *CA by iFish and normal LDH) | X | XX.X |
| II (Not R-ISS stage or III) | | |
| III(ISS stage III and either high-risk *CA by iFISH or high LDH) | | |
| Total | | |

<sup>(\*)</sup> Standard-risk (or standard prognosis) and high-risk as defined below

### 11.1.3 Cytogenetics

Table 11.1.3.1 Cytogenetics.

| Result ** | N | % |
|----------------|---|------|
| del13<br>del17 | X | XX.X |
| del17 | | |
| t(14;16) | | |
| Other* Total | | |
| Total | | |

Other (\*) Specify, see Listing 11.1.3.2

Listing 11.1.3.2 Cytogenetics: Result, 'Other'.

| Patient id. | Other |
|-------------|-------|

Patients will be classified in "high risk" or "standard prognosis" according to their genetic results (cytogenetic or FISH) at diagnosis or study entry.

Patients with translocations such as t(4;14), t(14;16), t(14;20), del 17, del 13 or single alterations such as +1q or +1p will be classified as "high risk"; patients with translocations such as t(11;14), t(6;14) or single alterations of trisomies 3, 5, 6, 9, 11, 15, 19 or 21 will be classified as "standard prognosis". This classification will be done by clinical review.

Table 11.1.3.3 Cytogenetic Risk.

| | N | % |
|---------------|---|------|
| Highrisk | X | XX.X |
| Standard risk | | |
| Total | | |

### 11.1.4 Prior Anticancer Therapy

Table 11.1.4.1 Number of Lines of Prior Medical Therapy.

| Two is 11.11. In 1 (while of of 2 most of 1 most with the way). | | |
|---|---|---|
| | N | % |
| 1 | X | XX.X |
| 2 | | |
| Total | | |
| Median (Range) | | |
| Mean (Std) | | |

N % CR sCR VGPR PR NE / NA / UNK Table 11.1.4.6 Status to Last Therapy Ν % Relapse Refractory Relapse/Refractory 11.1.5 Physical Examination, Vital Signs, Electrocardiogram and Other Tests For the physical examination, vital signs, electrocardiogram and other tests, the last examination available before or on treatment will be described in the following tables. Table 11.1.5.1 Baseline characteristics: Physical Exam. Parameter Median Mean StD Min Max Weight (kg.) Height (cm.) BSA (m<sup>2</sup>) Table 11.1.5.2 Number of Lesions (Plasmacytomas) at Baseline. No.of lesion % 1 lesion X 2 lesions 3 lesions See listing 11.1.5.3 for details 20 of 46

Median

%

XX.X

 $X\overline{X}.\overline{X}$ 

Min

Max

StD

X

N

Χ

Table 11.1.4.2 Prior Anti-myeloma Agents

Table 11.1.4.3 Prior Stem Cell Transplantation

Table 11.1.4.5 Best Response to Last Therapy

Median (Range) Mean (Std)

Autologous HSCT

Allogeneic HSCT

Time to progression. Last

anticancer therapy (months)

Both Total

Total

(ATC-level)

Table 11.1.4.4 TTP to Last Prior Anti-myeloma Therapy

Listing 11.1.5.3 Plasmacytomas at Baseline

| | Ĭ | New | Anatomic | Date | Method. | Lesion | Lesion | Product | Sum of |
|---|---|---|---|---|---|---|---|---|---|
| | | lesion | Localization | | | dim 1 | dim 2 | of the | the |
| Patient | T NI l | | | | | | | Cross- | product |
| id. | Lesion Number | | | | | | | diameters | of the |
| | | | | | | | | | Cross- |
| | | | | | | | | | Diameters |

Table 11.1.5.4 Baseline characteristics: Vital Signs.

| Parameter | N | Median | Mean | StD | Min | Max |
|---------------------------------|---|--------|------|-----|-----|-----|
| Heart rate (beats/min) | | | | | | |
| Systolic blood pressure (mmHg) | | | | | | |
| Diastolic blood pressure (mmHg) | | | | | | |
| Temperature (°C) | | | | | | |

Table 11.1.5.5 Baseline characteristics: Electrocardiogram

| | N | % |
|-------------------------------|---|------|
| Normal | X | XX.X |
| Significant abnormalities* | | |
| Non-significant abnormalities | | |
| Total | | |

<sup>(\*)</sup>See listing 11.1.5.6 for details

Listing 11.1.5.6 ECG Abnormalities at Baseline

| Patient id. | Result | QT interval (msec) | PR interval (msec) | QRS complex duration (msec) | Max Height of QRS (mm) | Heart Rate: | QTc (msec) |
|---|---|---|---|---|---|---|---|

### Table 11.1.5.7 Baseline Characteristics: ECOG Performance Status

| | N | % |
|-------|---|------|
| 0 | X | XX.X |
| 1 | | |
| 2 | | |
| Total | | |

### Table 11.1.5.8 Baseline characteristics: Neurological Examination

| | N | % |
|-----------|---|------|
| Normal | X | XX.X |
| Abnormal* | | |
| Total | | |

<sup>(\*)</sup>See listing 11.1.5.9 for details

### Listing 11.1.5.9 Neurological Examination Abnormalities at Baseline

| Patient id. | Result | Specify |
|-------------|--------|---------|

### Table 11.1.5.10 Baseline characteristics: LVEF

| | N | 0/0 |
|--------------------------------|---|------|
| Normal | X | XX.X |
| Significant abnormalities* | | |
| Non-significant abnormalities* | | |
| Total | | |

<sup>(\*)</sup>See listing 11.1.5.11 for details

Listing 11.1.5.11 Patients with Left Ventricular Ejection Fraction Abnormalities at Baseline

| Patient id. | Date | Method | LVEF (%) | Institutional normal range (%) | Result | Abnormalities |
|---|---|---|---|---|---|---|

### Table 11.1.5.12 Baseline Characteristics: Adequate Contraception

| | N | % |
|-------|---|------|
| Yes | X | XX.X |
| No | | |
| NA* | | |
| Total | | |

<sup>(\*)</sup> Specify reasons

Table 11.1.5.13 Baseline Characteristics: Pregnancy test

| | N | % |
|-----------------|---|------|
| Positive | X | XX.X |
| Negative<br>NA* | | |
| NA* | | |
| Not done | | |
| Total | | |

<sup>(\*)</sup> Specify reasons

### 11.1.6 Viral Serology

### Table 11.1.6.1 Viral Serology

| Two in the services | N | % |
|---------------------------------------|----|------|
| Viral caralagy | 1N | 70 |
| Viral serology | v | VVV |
| Yes | X | XX.X |
| Hepatitis B (HBC) | | |
| Surface antigen (HBsAg) | | |
| Positive | | |
| Negative | | |
| Not Done | | |
| Surface antibody (HBsAb or Anti-HBs): | | |
| Positive | | |
| Negative | | |
| Not Done | | |
| Core antibody (HBcAb or anti-HBc): | | |
| Positive | | |
| Negative | | |
| Not Done | | |
| Hepatitis C (HCV) | | |
| HCV | | |
| Positive | | |
| Negative | | |
| Not Done | | |
| Cytomegalovirus | | |
| CMV pp65 antigen | | |
| Positive | | |
| Negative | | |
| Not Done | | |
| Quantitative CMV DNA PCR | | |
| Positive | | |
| Negative | | |
| Not Done | | |

### 11.1.7 Hematological Values at Baseline

Table 11.1.7.1 Hematological Abnormalities at Baseline

| | N | Gı | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|------------------|---|----|----------|--------|----------|---|-----|
| | N | N | % | <br>N | % | N | % |
| Leukopenia | | | | | | | |
| Anemia | | | | | | | |
| Thrombocytopenia | | | | | | | |
| Neutropenia | | | | | | | |
| Lymphopenia | | | | | | | |

<sup>(\*)</sup>Any grade

Listing 11.1.7.2 Hematological Tests not Assessed at Baseline

| I | Patient id. | Lab. test |
|---|-------------|-----------|

Listing 11.1.7.3 Hematological Abnormalities at Baseline. Grade  $\geq 2$ 

| Patient id | Parameter | Value | Grade |
|------------|-----------|-------|-------|

#### 11.1.8 Biochemical Values at Baseline

Table 11.1.8.1 Biochemical Abnormalities at Baseline

| | N | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|--------------------------|---|----|----------|--------|----------|---|-----|
| | N | N | % | <br>N | % | N | % |
| AST increase | | | | | | | |
| ALT increase | | | | | | | |
| Total bilirubin increase | | | | | | | |
| AP increase | | | | | | | |
| Creatinine increase | | | | | | | |
| CPK increase | | | | | | | |
| GGT increase | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.8.2 Biochemical Values at Baseline

| | N | % |
|----------------------|---|---|
| LDH > 2 .5× ULN | | |
| B2-microglobulin>ULN | | |

Listing 11.1.8.3 Biochemical Tests not Assessed at Baseline

| Patient id. | Lab. test |
|-------------|-----------|

Listing 11.1.8.4 Biochemical Abnormalities at Baseline. Grade > 2

| Bisting 11:1:0.1 Bioenemical 1 tonormanties at Basenne. Grade _ 2 | | |
|---|---|---|
| Parameter | Value | Grade |

### 11.1.9 Other Metabolic Values at Baseline

Table 11.1.9.1 Other Metabolic Abnormalities at Baseline

| | N | Gr | ade<br>1 | <br>Gra | ade<br>4 | A | 11* |
|-----------------|---|----|----------|---------|----------|---|-----|
| | N | N | % | <br>N | % | N | % |
| Hyperglycemia | | | | | | | |
| Hypoglycemia | | | | | | | |
| Hypoalbuminemia | | | | | | | |

<sup>(\*)</sup>Any grade

Listing 11.1.9.2 Metabolic Tests not Assessed at Baseline

| Patient id. | Lab. test |
|-------------|-----------|

Listing 11.1.9.3 Metabolic Abnormalities at Baseline. Grade  $\geq 2$ 

| Patient id | Parameter | Value | Grade |
|------------|-----------|-------|-------|

### 11.1.10 Signs and Symptoms at Baseline

Table 11.1.10.1 Patients with Signs and Symptoms at Baseline

| | N | % |
|------------------------------------|---|---|
| No. signs and symptoms per patient | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (Range) | | |
| Mean (Std) | | |

Table 11.1.10.2 Signs and Symptoms at Baseline

| | | N | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | | N | % | <br>N | % | N | % |
| Gastrointestinal disorders | Diarrhea NOS | | | | | | | |
| | ••• | | | | | | | |
| General disorders and | Fatigue | | | | | | | |
| administration site conditions | ••• | | | | | | | |

<sup>(\*)</sup>Any grade

Listing 11.1.10.3 Signs and Symptoms at Baseline

| Eleving Tittote 2 | orgrin wire syrripterins at san | , • 11111• | | |
|---|---|---|---|---|
| Patient id. | Sign/symptom | Grade | Onset date | Treated |

### 11.1.11 Concomitant Medication/Procedures at Baseline

Concomitant medication at baseline according to the ATC classification.

Table 11.1.11.1 Agents of Concomitant Medication started at Baseline

| Medication Term (ATC level 1) | Medication Term<br>(ATC level 2) | Medication Term<br>(ATC level 4) | Preferred Name | N | % |
|---|---|---|---|---|---|
| | | | | X | XX.X |

Listing 11.1.11.2 Concomitant Medication Therapy at Baseline

| Patient id. | Туре | Drug name<br>/Procedure | ATC<br>Code | Route | Dose | Start date | End date | Ongoing | Indication |
|---|---|---|---|---|---|---|---|---|---|

Listing 11.1.11.3 Concomitant Procedures Therapy at Baseline

| Patient id. | Test | Date | Result |
|-------------|------|------|--------|

### 11.2 Efficacy Analysis

Efficacy analysis will be carried out on the "All Evaluable for Efficacy Patients" population.

### 11.2.1 Primary Analysis

Table 11.2.1.1 Overall Response

| Response | | |
|----------|---|---|
| | N | % |
| sCR | | |
| CR | | |
| VGPR | | |
| PR | | |
| MR | | |
| SD | | |
| PD | | |

Table 11.2.1.2 Overall Response Rate

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------------|------------|-----------------|-----------------|
| Response rate | | | |

Binomial exact estimator and 95% confidence interval

### 11.2.2 Secondary Analyses

Table 11.2.2.1 Duration of Response

| N |
|-----------|
| Events |
| Censored |
| Median DR |

Kaplan-Meier plot will be also shown (Figure 11.2.2.1)

Table 11.2.2.2 Time-To-Progression

| N |
|------------------|
| Events |
| Censored |
| Median TTP |
| TTP at 3 months |
| TTP at 6 months |
| TTP at 12 months |

Kaplan-Meier plot will be also shown (Figure 11.2.2.2)

Table 11.2.2.3 Progression-Free Survival

| N |
|------------------|
| Events |
| Censored |
| Median PFS |
| PFS at 3months |
| PFS at 6 months |
| PFS at 12 months |

Kaplan-Meier plot will be also shown (Figure 11.2.2.3)

#### Table 11.2.2.4 Event-Free Survival

| N |
|------------------|
| Events |
| Censored |
| Median EFS |
| EFS at 3 months |
| EFS at 6 months |
| EFS at 12 months |

Kaplan-Meier plot will be also shown (Figure 11.2.2.4)

#### Table 11.2.2.5 OS

| N |
|-----------------|
| Events |
| Censored |
| Median OS |
| OS at 6 months |
| OS at 12 months |

Kaplan-Meier plot will be also shown (Figure 11.2.2.5).

### 11.2.3 Other Exploratory Analyses

### Table 11.2.3.1 Clinical Benefit Rate

| | Proportion | Lower 95% limit | Upper 95% limit |
|-----------------------|------------|-----------------|-----------------|
| Clinical Benefit Rate | | | |

Binomial exact estimator and 95% confidence interval.

CBR defined as MR or better according to IMWG.

#### Table 11.2.3.2 Disease Control Rate

| | Proportion | Lower 95% limit | Upper 95% limit |
|----------------------|------------|-----------------|-----------------|
| Disease Control Rate | | | |

Binomial exact estimator and 95% confidence interval.

DCR defined as SD or better according to IMWG.

### Table 11.2.3.3 Duration of Minor Response

| N |
|-----------------------------------|
| Events |
| Censored |
| Median Duration of Minor Response |

Kaplan-Meier plot will be also shown (Figure 11.2.3.3)

### Table 11.2.3.4 Time to Response

| Twell III. |
|-------------------------------------|
| N |
| Events |
| Censored |
| Median Duration of Time to Response |

Kaplan-Meier plot will be also shown (Figure 11.2.3.4)

### 11.2.4 Characteristics of Responders

A summary of the main characteristics of patients with sCR, CR, VGPR, PR, MR or SD as best response will be shown.

Listing 11.2.4.1 Characteristics of Responders

| Patient id. | Sex | Age | PS | MM<br>type | Relapse<br>/Refractory | No. of prior lines | Cycles received | Best<br>response | PFS | DOR | <br>os |
|---|---|---|---|---|---|---|---|---|---|---|---|

### 11.2.5 Multivariate analyses

Multivariate analyses could be carried out as supportive analysis.

Table 11.2.5.1 Multivariate analysis of ORR

| Analysis of Maximum Likelihood Estimates | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates will be provided by the medical responsible

Table 11.2.5.2 Multivariate analysis of TTP

| | | | Analysis of M | laximum Like | elihood Est | imates | |
|---|---|---|---|---|---|---|---|
| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-<br>square | D 61:6 | 95% Hazard ratio confidence limits |

List of covariates will be provided by the medical responsible

Table 11.2.5.3 Multivariate analysis of PFS

| | | | Analysis of M | laximum Like | elihood Esti | mates | |
|---|---|---|---|---|---|---|---|
| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-square | Pr > ChiSq | 95% Hazard ratio confidence limits |

List of covariates will be provided by the medical responsible

Table 11.2.5.4 Multivariate analysis of EFS

| | Analysis of Maximum Likelihood Estimates | | | | | | |
|---|---|---|---|---|---|---|---|
| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-<br>square | Pr > ChiSq | 95% Hazard ratio confidence limits |

List of covariates will be provided by the medical responsible

Table 11.2.5.5 Multivariate analysis of OS

| | Analysis of Maximum Likelihood Estimates | | | | | | |
|---|---|---|---|---|---|---|---|
| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-<br>square | Pr > ChiSq | 95% Hazard ratio confidence limits |

List of covariates will be provided by the medical responsible

Figure 11.2.5.6. Response to Treatment per Cycle in All Patients Evaluable for Efficacy




### 12 Safety Analysis

Safety analysis will be carried out on the "All Evaluable for Safety Patients" population.

### 12.1 Extent of Exposure

### 12.1.1 Treatment Administration

Table 12.1.1.1 Number of Cycles Administered and Dose Intensity

| No. of cycles administered per patient | N | % |
|-----------------------------------------|---|---|
| 1 | | |
| 2 | | |
| 3 | | |
| Median (Range) | | |
| Mean (Std) | | |
| Time on treatment (weeks) | | |
| Median (Range) | | |
| Mean (Std) | | |
| Plitidepsin cumulative dose (mg/m²) | | |
| Median (Range) | | |
| Mean (Std) | | |
| Plitidepsin dose intensity (mg/m²/wk) | | |
| Median (Range) | | |
| Mean (Std) | | |
| Plitidepsin relative dose intensity (%) | | |
| Median (Range) | | |
| Bortezomib cumulative dose (mg/m²) | | |
| Median (Range) | | |
| Mean (Std) | | |
| Dexa cumulative dose (mg) | | |
| Median (Range) | | |
| Mean (Std) | | |

### 12.1.2 Cycle Delays

### 12.1.2.1 Number of Patients and Cycles with Dosing Delay, Any Relationship

Listing 12.1.2.1.1 Delays

| 215 11118 | | | , 5 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient id. | Cycle | Day | Previous cycle | Previous cycle start date | Delayed cycle | Delayed<br>cycle start<br>date | Dose Delay<br>calculated<br>(days) | Reason<br>for dose<br>delay | Dose<br>Delay<br>Spec. |

Table 12.1.2.1.2 Number of Patients and Cycles with Dosing Delay, any Relationship

| | N | % |
|-------------------------------------------|---|---|
| No. of patients susceptible of dose delay | | |
| No. of patients with any dose delay | | |
| No. of cycles administered | | |
| No. of cycles susceptible to be delayed* | | |
| No. of cycles with dosing delay** | | |
| No. of patients with | | |
| No plitidepsin delays | | |
| 1 cycle with plitidepsin delayed | | |
| 2 cycles with plitidepsin delayed | | |
| ≥ 3 cycles with plitidepsin delayed | | |
| No BTZ delays | | |

BTZ, bortezomib (\*) All cycles excluding first cycle. (\*\*) Denominator= Number of cycles susceptible to be delayed

Table 12.1.2.1.3 Number of Patients and Cycles with Dosing Delay according to the Relationship

| | Drug Related AE* | | Non-Drug Related<br>AE* | | Relationship<br>Unknown* | | Other* | |
|---|---|---|---|---|---|---|---|---|
| | N | % | N | % | N | % | N | % |
| No. of patients with 1 cycle delayed 2 cycles delayed ≥ 3 cycles delayed | | | | | | | | |
| No. of cycles with dosing delay* | | | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed.

Table 12.1.2.1.4 Length of Dosing Delay.

| | <u>C</u> | Treatmen | t-related** | Non-treatme | Total | | |
|---|---|---|---|---|---|---|---|
| Length of delay | Median (Range)<br>/Mean(Std) | | | | | | |
| Length of delay | | N | % | N | % | N | % |
| <= 7 days | <= 7 days | | | | | | |
| >7 days and <=14 days | | | | | | | |
| > 14 days | | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed. .(\*\*) Drug Related AE, Relationship unknown (\*\*\*)Non-drug related AE, other

### 12.1.2.2 Number of Delays according to Cycle Number

Listing 12.1.2.2.1 Cycle Delays due to AEs

| Patient id. | Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Resolved date | Significant consequences |
|---|---|---|---|---|---|---|---|---|

AEs with action = 'Dose delayed' or 'Dose delayed/reduced' or 'Dose delayed/omitted' or 'Dose de

#### 12.1.3 Dose Omissions

### 12.1.3.1 Number of Patients and Cycles with Dose Omissions

Listing 12.1.3.1.1 Dose Omissions

| Patient id. | | Cycle | Day | C | Cycle start date | Reason | n for dose<br>on | Dose omission Spec. |
|---|---|---|---|---|---|---|---|---|
| Listing 12.1.3.1.2 Dose Omissions due to AEs | | | | | | | | |
| Patient id. C | Cycle | Preferred term code | Adverse event reported | Grade | Relationship | Onset date | Resolved date | Significant consequences |

AEs with action = 'Dose Omitted' or 'Dose delayed/omitted' or 'Dose omitted/reduced' or 'Dose delayed/omitted/reduced'

#### 12.1.4 Dose Reductions

All dose reductions should be considered and described, specifying the reason for reduction (drug related AE, non-drug related AE, relationship unknown and other).

Listing 12.1.4.1 Dose Reductions

| Patient id. | Cycle | Day | Cycle start date | Previous dose | Reduced dose | Reason for dose reduction | Dose reduction Spec. |
|---|---|---|---|---|---|---|---|

Table 12.1.4.2 Number of Patients and Cycles with Dose Reduction, any Relationship

| | N | % |
|---|---|---|
| No. of patients treated | X | XX.X |
| No. of patients with any dose reduced | | |
| No. of patients with: | | |
| No plitidepsin reduction | | |
| 1 cycle with plitidepsin dose reduced | | |
| 2 cycles with plitidepsin dose reduced | | |
| No. of cycles administered | | |
| No. of cycles susceptible to have any dose reduced* | | |
| No. of cycles with plitidepsin dose reduced ** | | |
| No. of cycles with plitidepsin dose reduced (Treatment-related) ** | | |

<sup>(\*)</sup> All cycles excluding first cycle of those patients who have only received the first infusion. (\*\*) Denominator= Number of cycles susceptible to have a dose reduction

Table 12.1.4.3 Number of Patients and Cycles with Dose Reduction according to the Relationship

| Relationship | | |
|-------------------------------------|---|------|
| No. of cycles with dose reductions* | N | % |
| Treatment-related | | |
| Drug Related AE | X | XX.X |
| Relationship Unknown | | |
| Non-treatment-related | | |
| Non-Drug Related AE | | |
| Other * | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to have a dose reduction

Listing 12.1.4.4 Dose Reductions due to AEs

| Patient id. | Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Resolved<br>date | Significant consequences |
|---|---|---|---|---|---|---|---|---|

AEs with action = 'Dose Reduced' or 'Dose delayed/reduced or 'Dose omitted/reduced' or 'Dose delayed/omitted/reduced'

### 12.2 Adverse Events (AEs)

### 12.2.1 Display of Adverse Events

Table 12.2.1.1 Summary of Adverse Events.

| Table 12.2.1.1 Summary of Adverse Events. | N (%) |
|---|---|
| Patients with at least one AE regardless relationship | IN (70) |
| Any treatment-related AE | |
| Any plitidpesin-related AE | |
| Any BTZ -related AE | |
| Any DXM -related AE | |
| Any plitidepsin and DXM –related AE | |
| Any plitidepsin and BTZ –related AE | |
| Any DXM and BTZ –related AE Any DXM and BTZ –related AE | |
| Any phitidepsin&DXM&BTZ –related AE | |
| Any grade 3/4 AE | |
| Any grade 3/4 treatment-related AE | |
| Any grade 3/4 plitidpesin -related AE | |
| Any grade 3/4 BTZ -related AE Any grade 3/4 BTZ -related AE | |
| Any grade 3/4 DXM -related AE Any grade 3/4 DXM -related AE | |
| Any grade 3/4 plitidepsin and DXM –related AE | |
| Any grade 3/4 phitidepsin and BTZ –related AE Any grade 3/4 plitidepsin and BTZ –related AE | |
| Any grade 3/4 DXM and BTZ –related AE | |
| Any grade 3/4 plitidepsin&DXM&BTZ –related AE AEs leading to death | |
| AEs treatment-related leading to death | |
| AEs plitidpesin -related leading to death | |
| AEs BTZ -related leading to death | |
| AEs DXM -related leading to death | |
| AEs plitidepsin and DXM -related leading to death | |
| AEs plitidepsin and BTZ -related leading to death | |
| AEs DXM and BTZ -related leading to death | |
| AEs plitidepsin&DXM&BTZ -related leading to death | |
| AEs leading to dose delay | |
| AE treatment-related leading to dose delay | |
| AE plitidpesin -related leading to dose delay | |
| AE BTZ -related leading to dose delay | |
| AE DXM -related leading to dose delay | |
| AE plitidepsin and DXM -related leading to dose delay | |
| AE plitidepsin and BTZ -related leading to dose delay | |
| AE DXM and BTZ -related leading to dose delay | |
| AE plitidepsin&DXM&BTZ -related leading to dose delay | |
| AEs leading to dose omission | |
| AEs treatment-related leading to dose omission | |

| | N (%) |
|---|---|
| AEs plitidpesin -related leading to dose omission | |
| AEs BTZ -related leading to dose omission | |
| AEs DXM -related leading to dose omission | |
| AEs plitidepsin and DXM -related leading to dose omission | |
| AEs plitidepsin and BTZ -related leading to dose omission | |
| AEs DXM and BTZ -related leading to dose omission | |
| AEs plitidepsin&DXM&BTZ -related leading to dose omission | |
| AEs leading to treatment discontinuation | |
| AEs treatment-related leading to treatment discontinuation | |
| AEs plitidpesin -related leading to treatment discontinuation | |
| AEs BTZ -related leading to treatment discontinuation | |
| AEs DXM -related leading to treatment discontinuation | |
| AEs plitidepsin and DXM -related leading to treatment discontinuation | |
| AEs plitidepsin and BTZ -related leading to treatment discontinuation | |
| AEs DXM and BTZ -related leading to treatment discontinuation | |
| AEs plitidepsin&DXM&BTZ -related leading to treatment discontinuation | |
| AEs treatment-related leading to dose reduction | |
| AEs plitidpesin -related leading to dose reduction | |
| AEs BTZ -related leading to dose reduction | |
| AEs DXM -related leading to dose reduction | |
| AEs plitidepsin and DXM -related leading to dose reduction | |
| AEs plitidepsin and BTZ -related leading to dose reduction | |
| AEs DXM and BTZ -related leading to dose reduction | |
| AEs plitidepsin&DXM&BTZ -related leading to dose reduction | |

BTZ, bortezomib; DXM, dexamethasone

Table 12.2.1.2 Summary of Main Adverse Events.

| Main Adverse Events* | N (%) |
|------------------------------------|-------|
| Fatigue | |
| Diarrhea | |
| Peripheral Neuropathy | |
| Alanine aminotransferase increased | |

<sup>\*</sup> Main AEs will be defined by medical responsible (or will be defined as the most common AEs)

Table 12.2.1.3 Treatment-related\* Adverse Events. Worst Grade by Patient

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic<br>system disorders | Anemia NOS | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> or Unknown relationship (\*\*) Any grade

Table 12.2.1.4 Treatment-related\* Adverse Events. Worst Grade by Cycle

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic | Anemia NOS | | | | | | |
| system disorders | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> or Unknown relationship (\*\*) Any grade

Table 12.2.1.5 Adverse Events regardless of Relationship. Worst Grade by Patient

| | | | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic<br>system disorders | Anemia NOS | | | | | | |
| Cardiac disorders | <u>Arrhythmia NOS</u> | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.1.6 Adverse Events regardless of Relationship. Worst Grade by Cycle

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic<br>system disorders | Anemia NOS | | | | | | |
| Cardiac disorders | <u>Arrhythmia NOS</u> | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.1.7 Treatment Emergent Adverse Events\* .Worst Grade by Patient

| | | Gr | ade<br>1 | ••• | Gr | ade<br>4 | Al | 1** |
|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | | N | % | N | % |
| Blood and lymphatic<br>system disorders | Anemia NOS | | | | | | | |
| Cardiac disorders | <u>Arrhythmia NOS</u> | | | | | | | |
| | ••• | | | | | | | |

<sup>(\*)</sup>Treatment Emergent AE: Event that first appears during treatment, which was absent before or which worsens relative to the pre-treatment state (\*\*) Any grade

Table 12.2.1.8 Treatment Emergent Adverse Events. Worst Grade by Cycle

| | , -, | | | | | | |
|---|---|---|---|---|---|---|---|
| | | Gr | ade<br>1 | Gr | ade<br>4 | A | 11* |
| SOC | Preferred Term | N | % | N | % | N | % |
| Blood and lymphatic | Anemia NOS | | | | | | |
| system disorders | | - | | | | | |
| | ••• | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.2.1.9 Treatment-related\* Grade 3-4 Adverse Events. Worst Grade by Patient

| Patient id. | SOC Name | Preferred term | Grade |
|-------------|----------|----------------|-------|

<sup>(\*)</sup> or Unknown relationship (\*\*) Any grade

Listing 12.2.1.10 Treatment-related\* Grade 3-4 Adverse Events. Worst Grade by Cycle

| | | | | <u> </u> |
|-------------|-------|----------|----------------|----------|
| Patient id. | Cycle | SOC Name | Preferred term | Grade |

<sup>(\*)</sup> or Unknown relationship (\*\*) Any grade

Listing 12.2.1.11 Adverse Events Grade 3-4 regardless of Relationship. Worst Grade by Patient

| Patient id. | SOC Name | Preferred term | Grade |
|-------------|----------|----------------|-------|

# Listing 12.2.1.12 Adverse Events Grade 3-4 regardless of Relationship. Worst Grade by Cycle

| Patient id. | Cycle | SOC Name | Preferred term | Grade |
|-------------|-------|----------|----------------|-------|

At the time of the analysis, if appropriate, grouping of similar or clinically related items will be made.

### 12.3 Serious Adverse Events and deaths.

### 12.3.1 Serious Adverse Events

Table 12.3.1.1 Summary of Serious Adverse Events.

| , and the second | N (%) |
|---|---|
| Patients | |
| Any SAE | |
| Any treatment-related* SAE | |
| Any grade 3/4 SAE | |
| Any grade 3/4 treatment-related* SAE | |

<sup>(\*)</sup>Broken down by drug/drugs

Table 12.3.1.2 Treatment-related\* SAEs. Worst Grade by Patient

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic<br>system disorders | Anemia NOS | | | | | | |
| Cardiac disorders | <u>Arrhythmia NOS</u> | | | | | | |

<sup>(\*)</sup> or Unknown relationship (\*\*) Any grade

Table 12.3.1.3 Treatment-related\* SAEs. Worst Grade by Cycle

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic<br>system disorders | Anemia NOS | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> or Unknown relationship (\*\*) Any grade

Table 12.3.1.4 SAEs Regardless of Relationship. Worst Grade by Patient

| | | Gı | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic<br>system disorders | Anemia NOS | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.3.1.5 SAEs Regardless of Relationship. Worst Grade by Cycle

| 14010 12.5.1.5 5112 | b regulations of rectamen | bilip. Trois | Claa | $\mathbf{c}_{j}$ | , 010 | | | |
|---|---|---|---|---|---|---|---|---|
| | | Gı | ade<br>1 | | Gr | ade<br>4 | A | .11* |
| SOC | Preferred Term | N | % | | N | % | N | % |
| Blood and lymphatic<br>system disorders | Anemia NOS | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | |

<sup>(\*)</sup> Any grade

### Listing 12.3.1.6 SAEs

| Patient id. | Cycle | Preferred<br>term code | Adverse<br>event<br>reported<br>(verbatim) | Status | Grade | Relationship | Onset date | Resolved date | Action | Serious Criteria |
|---|---|---|---|---|---|---|---|---|---|---|

SAEs narratives will be provided by the pharmacovigilance department.

### 12.3.2 Deaths

### Table 12.3.2.1 Cause of Death

| Reason* | N | % |
|---------------------------|---|---|
| Malignant disease | | |
| Study drug related AE | | |
| Non study drug related AE | | |
| Other | | |
| Total | | |

<sup>(\*)</sup> Denominator=Number of patients who died.

### Listing 12.3.2.2 Deaths

| Patient id. | Death date | Cause | Autopsy | Autopsy report available | Number of cycles administered | Last infusion date | Time on treatment* | Time from<br>Last dose** |
|---|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>Time on treatment: defined as last infusion date plus 30 days, or date of death or subsequent therapy (whichever comes first) minus first infusion date. (\*\*)Time from last dose defined as death date minus last infusion date.

### Listing 12.3.2.3 Deaths due to AEs

| Patient id | . Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset date | Resolved date | Action |
|---|---|---|---|---|---|---|---|---|

### 12.4 Clinical laboratory evaluation

### 12.4.1 Hematological Abnormalities

Table 12.4.1.1 Hematological Abnormalities during Treatment, Worst Grade per Patient

| 3 | N Grade | | | Grade<br>4 | | All* | | |
|------------------|---------|---|----|------------|---|------|---|---|
| | N | N | % | | N | % | N | % |
| Anemia | | | | | | | | |
| Leukopenia | | | | | | | | |
| Neutropenia | | | | | | | | |
| Lymphopenia | | | | | | | | |
| Thrombocytopenia | | | Ţ, | · | | | | |

(\*) Any grade

Table 12.4.1.2 Hematological Abnormalities during treatment, Worst Grade per Cycle

| | N | Grade<br>1 | | ••• | Grade<br>4 | | All* | |
|------------------|---|------------|---|-----|------------|---|------|----|
| | N | N | % | | N | % | N | % |
| Anemia | | | | | | | | |
| Leukopenia | | | | | | | | |
| Neutropenia | | | | | | | | |
| Lymphopenia | | | | | | | | |
| Thrombocytopenia | | | | · | | | | Ţ, |

(\*) Any grade

Listing 12.4.1.3 Grade 3-4 hematological Abnormalities during Treatment. Worst Grade per Patient

| _ F | | |
|-------------|------|-------|
| Patient id. | Test | Grade |

Listing 12.4.1.4 Grade 3-4 hematological Abnormalities during Treatment. Worst Grade per Cycle

| Patient id. | Test | Grade |
|-------------|------|-------|

Listing 12.4.1.5 Hematological Tests not Assessed at any Treatment Visit per Patient

| | issessed at the property is to perform the performance of the performa |
|---|---|
| Patient id. | Lab. test |

Listing 12.4.1.6 Hematological Tests not Assessed by Patient and Cycle

| Patient id. | Cycle | Lab. test |
|-------------|-------|-----------|

Table 12.4.1.7 Blood Products during the study

| | N | % |
|------------------|---|------|
| Packed red cells | X | XX.X |
| Platelets | | |
| Plasma | | |
| Cryoprecipitates | | |
| Clotting factors | | |

These tables will be complemented with plots for the median nadir of neutrophils (Figure 12.4.1.8), platelets count (Figure 12.4.1.9) and hemoglobin values (Figure 12.4.1.10) by cycle along the treatment. Furthermore, if appropriate, graphs of the intercycle time course of neutropenia and thrombocytopenia will be provided.

#### 12.4.2 Biochemical Abnormalities

Table 12.4.2.1 Biochemical Abnormalities during Treatment, worst Grade per Patient

| | N | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|--------------------------|---|----|----------|--------|----------|---|-----|
| | N | N | % | <br>N | % | N | % |
| AST increase | | | | | | | |
| ALT increase | | | | | | | |
| Total bilirubin increase | | | | | | | |
| AP increase | | | | | | | |
| Creatinine increase | | | | | | | |
| CPK increase | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.4.2.2 Biochemical Abnormalities during Treatment, Worst Grade per Cycle

| | N | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|--------------------------|---|----|----------|--------|----------|---|-----|
| | N | N | % | <br>N | % | N | % |
| AST increase | | | | | | | |
| ALT increase | | | | | | | |
| Total bilirubin increase | | | | | | | |
| AP increase | | | | | | | |
| Creatinine increase | | | | | | | |
| CPK increase | | | | | | | |
| (4) 4 1 | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.2.3 Grade 3-4 biochemical Abnormalities during Treatment. Worst Grade per Patient

| Patient id. | Test | Grade |
|-------------|------|-------|

Listing 12.4.2.4 Grade 3-4 biochemical Abnormalities during Treatment. Worst Grade per Cycle

| Patient id. | Cycle | Test | Grade |
|-------------|-------|------|-------|

Listing 12.4.2.5 Biochemical tests not Assessed at any Treatment Visit by Patient

| | t diriy 11 comment + 1810 cy 1 deletic |
|-------------|----------------------------------------|
| Patient id. | Lab. test |

Listing 12.4.2.6 Biochemical Tests not Assessed by Patient and Cycle

| Datiant id | Consta | Lah test |
|-------------|--------|-----------|
| Patient id. | Cycle | Lab. test |

These tables will be complemented with plots for the median peak of ALT (Figure 12.4.2.7, AST (Figure 12.4.2.8) and CPK values (Figure 12.4.2.9) by cycle along the treatment. If appropriate, graphs of the intercycle time course of ALT, AST and CPK will be provided.

### 12.4.3 Other metabolic parameters

Table 12.4.3.1 Metabolic Abnormalities during Treatment, Worst Grade per Patient

| | N | Gı | rade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|-----------------|---|----|-----------|--------|----------|---|-----|
| | N | N | % | <br>N | % | N | % |
| Hyperglycemia | | | | | | | |
| Hypoglycemia | | | | | | | |
| Hypoalbuminemia | | | | | | | |

(\*) Any grade

Table 12.4.3.2 Metabolic Abnormalities during Treatment, Worst Grade per Cycle

| | N | Gr | ade<br>1 | <br>Gr | ade<br>1 | A | 11* |
|-----------------|---|----|----------|--------|----------|---|-----|
| | | N | % | <br>N | % | N | % |
| Hyperglycemia | | | | | | | |
| Hypoglycemia | | | | | | | |
| Hypoalbuminemia | | | | | | | |

(\*) Any grade

Listing 12.4.3.3 Grade 3-4 metabolic Abnormalities during Treatment. Worst Grade by Patient

| Patient id. | Test | Grade |
|-------------|------|-------|

Listing 12.4.3.4 Grade 3-4 metabolic Abnormalities during Treatment. Worst Grade by Cycle

| Patient id. | Cycle | Test | Grade |
|-------------|-------|------|-------|

Listing 12.4.3.5 Metabolic Tests not Assessed at any Treatment Visit by Patient

| Patient id. | Lab. test |
|-------------|-----------|

Listing 12.4.3.6 Metabolic Tests not Assessed by Patient and Cycle

| Patient id. | Cycle | Lab. test |
|-------------|-------|-----------|

### 12.4.4 Laboratory values over time

Table 12.4.4.1 Evolution of Hematological Abnormalities from Baseline, Worst Case per Patient.

| | | | | V | Vorst gr | ade per p | atient | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 0 | | 1 | | | Total | |
| | | | N | % | N | % | N | % | N | % |
| | Neutropenia | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| o o | Thrombocytopenia | | | | | | | | | |
| i | | Grade 0 | | | | | | | | |
| ase | | Grade 1 | | | | | | | | |
| Щ | | | | | | | | | | |
| | | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

Table 12.4.4.2 Worsening of Hematological Abnormalities from Baseline, Worst Case per Patient.

| | | | | V | Vorst gr | ade per p | atient | | т | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 0 | | 1 | | | 1 | otai |
| | | | N | % | N | % | N | % | N | % |
| | Neutropenia | Grade 0 | | | | | | | | |
| | Grad Thrombocytopenia Grad | Grade 1 | | | | | | | | |
| ine | | Grade 0 | | | | | | | | |
| sel | | Grade 1 | | | | | | | | |
| Ba | | | | | | | | | | |
| | •••• | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

Table 12.4.4.3 Evolution of Biochemical Abnormalities from Baseline, Worst Case per Patient.

| | | | | Worst grade per patient | | | | | | oto1 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 0 | | 1 | | | | Total |
| | | | N | % | N | % | N | % | N | % |
| | AST increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| ine | · <b>-</b> | Grade 0 | | | | | | | | |
| seli | | Grade 1 | | | | | | | | |
| Ba | | | | | | | | | | |
| | •••• | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | | ••••• | | | | | | | | |

Table 12.4.4.4 Worsening of Biochemical Abnormalities from Baseline, Worst Case per Patient.

| | | | | W | orst grad | le per pa | tient | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 0 | | 1 | | | Total | |
| | | | N | % | N | % | N | % | N | % |
| A | AST increase | Grade 0 | | | | | | | | |
| | ALT increase Grade 0 Grade 1 Grade 0 Grade 1 Grade 1 | Grade 1 | | | | | | | | |
| A B. | | Grade 0 | | | | | | | | |
| sel | | Grade 1 | | | | | | | | |
| Ba | | | | | | | | | | |
| | Gra | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

Table 12.4.4.5 Grade 3-4 laboratory Abnormalities in the First Cycle and in all Other Cycles

| Laboratory | | Cycle 1 | | Сус | le>1 | |
|---|---|---|---|---|---|---|
| abnormalities | No. of cycles evaluated No. of cycles grade 3-4 | | % | No. of cycles evaluated No. of cycle grade | | % |
| Thrombocytopenia | | | | | | |
| Neutropenia | | | | | | |
| AP | | | | | | |
| Total bilirubin | | | | | | |
| AST | | | | | | |
| ALT | | | | | | |
| СРК | | | | | | |

Table 12.4.4.6 ALT, AST and CPK Time-Course Pattern

| | Onset day<br>grade 3/4 | Days in grade 3/4 | Time to recovery to grade <=2 | | |
|---|---|---|---|---|---|
| Laboratory abnormalities | <i>3</i> | | Median | 95%CI<br>Lower limit | 95%CI<br>Upper limit |
| ALT | | | | | |
| AST | | | | | |
| СРК | | | | | |

If considered relevant CPK relationship with muscular toxicity will be studied by means of descriptive tables/listings.

Table 12.4.4.7 Platelet Count and Neutrophil Count Time-Course Pattern

| | Onset day grade 3/4 | Days in grade 3/4 | Time to | ade <=2 | |
|---|---|---|---|---|---|
| Laboratory abnormalities | | | Median | 95%CI<br>Lower limit | 95%CI<br>Upper limit |
| Platelet count | | | | | |
| Neutrophil count | | | | | |

### 12.5 Vital Signs, Physical Findings, LVEF, ECG and Other Tests Related to Safety

### 12.5.1 Vital Signs and Physical Findings

Table 12.5.1.1 ECOG Performance Status during the Study

| | | Cycle/PS* | | | |
|-------------|---|-----------|---|---|----|
| | 0 | 1 | 2 | 3 | •• |
| Patient id. | | | | | |

<sup>(\*)</sup> Worst ECOG PS of the cycle determinations.

Table 12.5.1.2 Physical Examination during the Study.

| | | Cycle/Physical examination result* |
|-------------|---|------------------------------------|
| | 0 | 0 1 2 3 4 |
| Patient id. | | |

<sup>(\*)</sup> Worst result per cycle.

### Table 12.5.1.3 Weight by Patient per Cycle

| | | Cycle/Weight | | |
|-------------|-----------|--------------|-----------|-----------|
| | 0<br>(kg) | 1*<br>(%) | 2*<br>(%) | 3*<br>(%) |
| Patient id. | | | | |

<sup>(\*) %</sup> of changes respect to baseline

Table 12.5.1.4 Number of Lesions (Plasmacytomas) during the Study.

| | | Cycle/No of lesions* | | | |
|-------------|---|----------------------|---|---|----|
| | 0 | 1 | 2 | 3 | •• |
| Patient id. | | | | | |

<sup>(\*)</sup>Max.number of lesions of the cycle determinations.

### 12.5.2 LVEF and ECG

Listing 12.5.2.1 LVEF Evolution during the Study

| Patient id. | LVEF(%) | | |
|---------------|-----------|----------|-------------------|
| i attent id. | Baseline* | Minimun* | End of treatment* |
| Median(Range) | | | |
| Mean(Std) | | | |

<sup>(\*)</sup> LVEF (%) value and method

Listing 12.5.2.2 Electrocardiogram Results . Evolution during the Study.

| Patient id. | Cycle | ECG result |
|-------------|-------|------------|

### 12.6 Concomitant Medication / Procedures according to the ATC Classification.

Table 12.6.1 Concomitant Medication during Treatment (ATC levels)

| | | | | <i>'</i> | |
|---|---|---|---|---|---|
| Medication Term | Medication Term | Medication Term | Preferred Name | | |
| (ATC level 1) | (ATC level 2) | (ATC level 4) | Preferred Name | N | % |
| | | | | X | XX.X |

Table 12.6.2 G-CSF, transfusions and Bisphosphonates during Treatment

| | N | % |
|-------|---|---|
| G-CSF | | |

| Table 12.6.3 Subsequent Therapy | | |
|---------------------------------|---|---|
| | N | % |
| Туре | | |

Table 12.6.4 Time to subsequent therapy or death

| N | X |
|-------------|-----|
| Events | X |
| Censored | X |
| Median Time | X.X |

Kaplan-Meier plot will be also shown (Figure 12.6.4)

Subsequent chemotherapy agents (ATC)

Chemotherapy

### 12.7 Safety Analysis in Special Subgroups.

Table 12.7.1 Worst grade 3-4 by patient in special subgroups (Race)

| | White | | | Other | | |
|------------------|-------|-----------|-----|-------|-----------|-----|
| | N | Grade 3-4 | % | N | Grade 3-4 | % |
| Thrombocytopenia | X | X | X.X | X | X | X.X |
| Neutropenia | | | | | | |
| AP | | | | | | |
| Total bilirubin | | | | | | |
| AST | | | | | | |
| ALT | | | | | | |
| СРК | | | | | | |
| Nausea | | | | | | |
| Vomiting | | | | | | |
| Fatigue | | | | | | |
| Other* | | | | | | |

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group

### 12.8 MM Serum/Urine Protein Measurements

Figure 12.8.1 Individual M-protein Values of Responder Patients



Figure 12.8.2 Waterfall Plot. (Maximum Reduction of M-Protein in Serum/Urine)

Maximal variation M-Protein



#### APPENDIX II

### 13 DB Listings

### CRF Listings.

-Listing 13.1.1: Screening -Listing 13.1.2: Demographics -Listing 13.1.3: Contraception/Pregnancy test -Listing 13.1.4: Medical history -Listing 13.1.5: MM history -Listing 13.1.6: Cytogenetics -Listing 13.1.7: Prior AntiCancer Therapy: Surgery -Listing 13.1.8: Prior AntiCancer Therapy: Palliative RadioTherapy -Listing 13.1.9: Prior AntiCancer Medical Therapy for Study Disease -Listing 13.1.10: Hematology laboratory values -Listing 13.1.11: Coagulation Test -Listing 13.1.12: Biochemical laboratory values -Listing 13.1.13: Other metabolic laboratory values -Listing 13.1.14: Urinalysis -Listing 13.1.15: Physical examination -Listing 13.1.16: Clinical neurological assessment -Listing 13.1.17: Performance status -Listing 13.1.18: Vital signs -Listing 13.1.19: Electrocardiogram -Listing 13.1.20: Left Ventricular Ejection Fraction -Listing 13.1.21: Viral Serology -Listing 13.1.22: Prophylactic medication -Listing 13.1.23: Oral Dexamethasone Administration -Listing 13.1.24: Plitidepsin Administration -Listing 13.1.25: Plitidepsin Readministration -Listing 13.1.26: Bortezomib Administration -Listing 13.1.27: Treatment Continuation -Listing 13.1.28: Adverse events (including signs and symptoms) -Listing 13.1.29: SAE Summary -Listing 13.1.30: Concomitant Medication/Procedures/Other Test -Listing 13.1.31: Blood products use -Listing 13.1.32: End of treatment -Listing 13.1.33: Unscheduled -Listing 13.1.34: Follow up -Listing 13.1.35: Radiotherapy (after End of Treatment) -Listing 13.1.36: Medical Treatment (after End of Treatment) -Listing 13.1.37: MM Serum Protein Measurements

-Listing 13.1.38: MM Urine Protein Measurements

-Listing 13.1.39: Disease Evaluation -Listing 13.1.40: C-Reactive Protein

- -Listing 13.1.41: Beta-2-microglobulin
- -Listing 13.1.42: Tumor Evaluation (Plasmacytomas)
- -Listing 13.1.43: Skeletal Evaluation
- -Listing 13.1.44: Bone Marrow Evaluation
- -Listing 13.1.45: Evaluation of Response
- -Listing 13.1.46: Death Report Form
- -Listing 13.1.47: Off Study

#### APPENDIX III

### 14 ICH Listings

In accordance with ICH E-3 guidelines, the patient listings specified as Section 16.2 will be prepared.

- 16.2.1 Discontinued Patients
- 16.2.2 Protocol Deviations
- 16.2.3 Patients Not Included in the Efficacy Analysis
- 16.2.4 Demographic Data
- 16.2.5 Compliance and/or Drug Concentration Data
- 16.2.6 Individual Efficacy Response Data
- 16.2.7 Adverse Event Listing (each patient)
- 16.2.8 Listing of Individual Laboratory Measurements by Patient